CLINICAL TRIAL: NCT00976651
Title: Influence of Ovarian Stimulation With 200 IU of hCG, (Administered in the Late Follicular Phase Among ICSI Patients Undergoing a GnRH-antagonist Protocol), on the Endometrium on the Day of Oocyte Pick-up
Brief Title: Low Dose Human Chorionic Gonadotropin: Influence on the Endometrium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Paul Devroey, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBLD2
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2009-09

CONDITIONS: Infertility
Keywords: infertility; ICSI; hCG; infertility treatment
MeSH Terms: conditions — Infertility | interventions — Menotropins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recombinant FSH (Active Comparator): Patients undergo a standard antagonist protocol for in-vitro fertilisation, and are stimulated with recombinant gonadotropins. Histology and gene expression is studied on the endometrium.
  Interventions: Drug: human menopausal gonadotropin
- human chorionic gonadotropin (Experimental): Patients undergo an antagonist protocol for in-vitro fertilisation and are stimulated with recombinant gonadotropins. When the patient has an estradiol value of 600 ng/L or more and when the patient has at least 6 follicles of 12 mm, the administration of gonadotropins is stopped and replaced by low dose human chorionic gonadotropins.
  Histology and gene expression is studied on the endometrium
  Interventions: Drug: human menopausal gonadotropin

INTERVENTIONS:
Drug: human menopausal gonadotropin — 200 IU per day in the late follicular phase

SUMMARY:
The purpose of the present study is to assess the influence of the administration of low dose hCG on the endometrium. The study is a randomised trial where 2 groups of patients, undergoing a gonadotropin-releasing hormone antagonist protocol for in vitro fertilization, are studied. In addition to the histological findings, by analysing the correlation of the morphological pattern and gene expression profile of human endometrium on the day of oocyte retrieval in patients of both treatment groups, the investigators want to study the implantation potential.

ELIGIBILITY:
Inclusion Criteria:

* < 36 years on day of randomisation
* FSH < 12 in the early follicular phase
* Normal ultrasound scan
* BMI between 18 and 29 (both inclusive)
* Randomisation at outpatient clinic

Exclusion Criteria:

* Endometriosis ≥ grade 3
* PCO syndrome
* Poor responder
* Endocrine or metabolic abnormalities

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
number of oocytes | 2 weeks after start of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Laarbeeklaan 101, Brussels Capital, Belgium

REFERENCES:
- [Result] Blockeel C, De Vos M, Verpoest W, Stoop D, Haentjens P, Devroey P. Can 200 IU of hCG replace recombinant FSH in the late follicular phase in a GnRH-antagonist cycle? A pilot study. Hum Reprod. 2009 Nov;24(11):2910-6. doi: 10.1093/humrep/dep253. Epub 2009 Jul 17. PMID 19617207